CLINICAL TRIAL: NCT05813938
Title: Assessment of Accuracy and Safety of LabTest Checker - Clinical Evaluation of a Patient-centered Clinical Decision Support System Based on AI
Brief Title: Assessment of Accuracy and Safety of LabTest Checker
Acronym: LTC-AI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Labplus Sp. z o.o. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LP001
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Abnormalities in the Blood Test Results
Keywords: laboratory test interpretation; artificial intelligence; clinical decision support system; clinical implementation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental)
  Interventions: Device: LabTest Checker

INTERVENTIONS:
Device: LabTest Checker — A set of blood laboratory tests is ordered. Test results are recorded in the LabTest Checker. LabTest Checker's diagnostic engine automatically generates a personalized questionnaire that is filled out by the patient. After obtaining all necessary information, including the patient's chronic diseases, medications taken, and symptoms, the tool presents an interpretation of test results.

SUMMARY:
The goal of this study is to assess performance of a new clinical decision support system named LabTest Checker in a cohort of adult patients reporting to the internal ward's emergency department. The main question it aims to answer is:

• how accurate and safe is LabTest Checker.

A set of blood laboratory tests will be ordered for each participant. Participants will use LabTest Checker to obtain an interpretation of their test results. The interpretation provided by LabTest Checker will then be compared with the interpretation given by an internal medicine specialist to assess the accuracy and safety of the tool.

ELIGIBILITY:
Inclusion Criteria:

* adult
* requires laboratory test investigation

Exclusion Criteria:

* under 18 years old
* pregnant
* no need for laboratory test investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
accuracy | 7 days
  the ratio of the number of patients for whom the LTC correctly assigned triage category to the total number of patients
sensivity to emergency | 7 days
  the ratio of the number of cases correctly identified as emergency by the LTC to the number of cases identified as emergency by the physician
sensivity to urgency | 7 days
  the ratio of the number of cases correctly identified as urgency by the LTC to the number of cases identified as urgency by the physician
safety | 7 days
  the ratio of the number of patients for whom a triage category assigned by the LTC was higher than or equal to the triage category assigned by the physician to the total number of cases

SECONDARY OUTCOMES:
reduction of unnecessary visits | 7 days
  the ratio of the number of patients who will avoid at least one unnecessary consultation by following the LabTest Checkers recommendations to the total number of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Oddział Chorób Wewnętrznych i Chemioterapii Onkologicznej, Samodzielny Publiczny Szpital Kliniczny im. Andrzeja Mielęckiego Śląskiego Uniwersytetu Medycznego w Katowicach, Katowice, Poland